CLINICAL TRIAL: NCT01622075
Title: A Multicenter, Randomized, Active Controlled Clinical Study to Evaluate the Safety and Efficacy of the Treatment of In-stent Restenosis Lesion by Paclitaxel-eluting PTCA- Balloon Catheter Versus Paclitaxel-eluting Stent
Brief Title: A Safety and Efficacy Study of Paclitaxel-eluting Balloon to Paclitaxel-eluting Stent
Acronym: PEPCAD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: B. Braun Medical International Trading Company Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AE-V-S-1001
Record Dates: First submitted 2012-06-05; First posted 2012-06-18 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Coronary Instent Restenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SeQuent® Please (Experimental): Paclitaxel Drug-eluting Coronary Artery Balloon Catheter
  Interventions: Device: SeQuent® Please
- Taxus Liberte (Active Comparator): Paclitaxel Drug-eluting Coronary Stent and Conveying System
  Interventions: Device: Taxus Liberte

INTERVENTIONS:
Device: SeQuent® Please — SeQuent® Please with a length of 10mm,15mm,17mm,20mm and 26mm and diameter of 2.5 mm, 2.75 mm, 3.0mm, 3.5mm and 4.0mm are to be used in the trial
  Other Names: Paclitaxel Drug-eluting Coronary Artery Balloon Catheter
  Arms: SeQuent® Please
Device: Taxus Liberte — Taxus Liberte with a length of 8mm,12mm,16mm,20mm and 24mm and diameter of 2.5 mm, 2.75 mm, 3.0mm, 3.5mm and 4.0mm are to be used in the trial
  Other Names: Paclitaxel Drug-eluting Coronary Stent and Conveying System
  Arms: Taxus Liberte

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of successful interventional therapy and unblocked blood vessel maintaining in the treatment of coronary in-stent restenosis by paclitaxel -eluting PTCA- balloon catheter (3μg/mm2 balloon surface area) versus paclitaxel-eluting stent Taxus® Liberte, and the reference diameter of coronary artery stenosis is 2.5mm-4.0mm and the length ≤30mm.

ELIGIBILITY:
Inclusion Criteria:

1. Related to patients

   * Patients with stable angina, unstable angina, old myocardial infarction or proven asymptomatic ischemia
   * Restenosis after the first stent implant
   * Patients who can receive any kind of coronary revascularization (including balloon angioplasty, stent implantation or coronary artery bypass grafting)
   * Patient aged 18-80 (including 18 and 80)
   * Female patients of childbearing age in the study period shall not be pregnant or protocol to be pregnant, it is suggested that patients shall take sufficient contraception measures till (including) the follow-up visit of month 9
   * Patients who agree to accept the angiography follow-up visits of month 9
   * Patients who agree to accept the clinical visits at Day 30, Month 6 and Month 12
   * Patients can understand the study objectives psychologically and linguistically and show the sufficient compliance to the study protocol. Patients present acceptance of the risks and benefits described in the informed consent form.
2. Related to lesion

   * Drug-eluting stent restenosis: Type Mehran I, Type II and Type III; the reference blood vessel diameter is 2.5 mm-4.0 mm, length ≤30mm
   * Before surgery, stenosis diameter must be ≥70% or ≥50% and accompanied by ischemia
   * The distance between other lesion requires interventional therapy and the target lesion must be >10mm
   * In the stent group, up to two paclitaxel drug stents are permitted to be implanted in series

Exclusion Criteria:

1. Related to patients

   * Patients with myocardial infarction within one week
   * Patients with severe congestive heart failure or NYHA IV severe heart failure
   * Patients with severe valvular heart disease
   * Female patients in pregnancy or lactation
   * Patients with the life expectancy not exceeding 1 year or the factors causing difficult clinical follow-up visits
   * Patients with hemorrhagic tendency, prohibited to take anticoagulants or antiplatelet drugs
   * Patients with stroke within 6 months before the surgery
   * Patients taking part in any other clinical tests
   * Existing sever renal failure (GFR<30ml/min) or the history, so not meeting the conditions of angiography
   * Patients with cardiac transplantation
   * Patients not included for other reasons from the investigators
2. Related to lesion

   * Evidence of extensive thrombus in target blood vessel before the intervention
   * Percutaneous coronary intervention for many in-stent restenosis lesions in same artery
   * 3-vessel disease that all need to be intervented
   * In bifurcation lesions, branch open blood vessel diameter ≥2.5mm
   * Percutaneous coronary intervention of venous graft
   * Entire shut of Grade TIMI 0 blood flow (Type Mehran IV stenosis)
   * Open lesion at left primary and within 2mm
3. Related to concomitant therapy

   * Patients cannot tolerate aspirin and/or clopidogrel, patients with the history of neutrocytopenia or thrombocytopenia, or patients with severe hypohepatia and prohibited to take clopidogrel
   * Patients known allergic to paclitaxel
   * Patients with the history of leucopenia (numeration of leukocytes <3x109/L, exceeding 3 days), neutrocytopenia (ANC<1000 neutrocytes/mm3, exceeding 3 days) or thrombocytopenia (<100,000 platelets/mm3
   * Patients with the history of peptic ulcer or gastrointestinal hemorrhage in the past 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2011-03; Primary Completion 2013-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Late lumen loss in segment section at M9 | One year
  To measure the diameter loss in segment restenosis of the target lesion vessel by using angiography

SECONDARY OUTCOMES:
Success rate of the interventional therapy | Two year
  To compare the successful treatment of coronary artery stent restenosis intervention between Paclitaxel release PTCA balloon and Taxus® Liberte, including apparatus success, lesion success and clinical success
Outcomes of clinical follow-up visits for drug stent versus drug balloon | Two year
  * Binary restenosis rate in lesion section at M9
  * Cardiovascular clinical composite endpoints related to apparatus at D30, M6, M9, M12 and M24, including cardiac death, target blood vessel myocardial infarction and target lesion vessel revascularization driven by clinical symptoms, briefed as target lesion failure
  * Cardiovascular clinical composite endpoints related to patients at D30, M6, M9, M12 and M24, including all-cause death, all myocardial infarction and any vessel revascularization
  * Thrombus event rate defined by ARC

CONTACTS AND LOCATIONS:
Overall Officials: Runlin Gao, Prof., Principal Investigator — Fuwai CVD Hospital of Chinese Academy of Medical Sciences
Locations (1):
- Fuwai CVD Hospital of Chinese Academy of Medical Sciences, Beijing, China

REFERENCES:
- [Derived] Xu B, Qian J, Ge J, Wang J, Chen F, Chen J, Wei M, Chen Y, Yang Y, Gao R; PEPCAD China ISR investigators. Two-year results and subgroup analyses of the PEPCAD China in-stent restenosis trial: A prospective, multicenter, randomized trial for the treatment of drug-eluting stent in-stent restenosis. Catheter Cardiovasc Interv. 2016 Mar;87 Suppl 1:624-9. doi: 10.1002/ccd.26401. Epub 2016 Jan 17. PMID 26775079
- [Derived] Xu B, Gao R, Wang J, Yang Y, Chen S, Liu B, Chen F, Li Z, Han Y, Fu G, Zhao Y, Ge J; PEPCAD China ISR Trial Investigators. A prospective, multicenter, randomized trial of paclitaxel-coated balloon versus paclitaxel-eluting stent for the treatment of drug-eluting stent in-stent restenosis: results from the PEPCAD China ISR trial. JACC Cardiovasc Interv. 2014 Feb;7(2):204-211. doi: 10.1016/j.jcin.2013.08.011. PMID 24556098